CLINICAL TRIAL: NCT06581094
Title: Effects of UC-II, Glucosamine and Curcumin Supplementation on Knee Pain and Inflammation: A Randomized, Single-blind, Placebo-controlled Parallel-group Trial
Brief Title: Effects of UC-II, Glucosamine and Curcumin Supplementation on Knee Pain and Inflammation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202406039
Record Dates: First submitted 2024-08-29; First posted 2024-09-03 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2024-07

CONDITIONS: Inflammation; Knee Pain Chronic
Keywords: Non-denatured type II collagen; Glucosamine; Curcumin; Knee Pain
MeSH Terms: conditions — Inflammation | interventions — Glucosamine; Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Control group use 42 mg UCII.
  Interventions: Dietary Supplement: Placebo
- Test group (UCII, glucosamine, and curcumin) (Experimental): Test group use 42 mg UCII, 460 mg glucosamine and 380 mg curcumin
  Interventions: Dietary Supplement: UCII, glucosamine and curcumin

INTERVENTIONS:
Dietary Supplement: UCII, glucosamine and curcumin — compound capsules twice daily.
  Arms: Test group (UCII, glucosamine, and curcumin)
Dietary Supplement: Placebo — Placebo capsules twice daily.
  Arms: Control group

SUMMARY:
This research evaluated the effects of UCII, glucosamine and curcumin supplementation on knee pain and inflammation.

DETAILED DESCRIPTION:
Arthritis is an inflammation of one or more joints, characterized by pain, stiffness (especially in the early morning or after exercise), swelling, deformation, and/or reduced mobility. There are many different forms of arthritis. Osteoarthritis, also known as degenerative arthritis, is caused by abnormal damage to the cartilage at the ends of bones. In some patients, it is caused by injury or congenital abnormalities in the proteins that make up cartilage. Generally, it seems that aging, an unbalanced diet, and an inappropriate lifestyle are the causes of this disease.

Once the cartilage tissue changes from smooth to rough or breaks into small pieces, the cartilage is gradually destroyed, and the normally smooth surface becomes irregular. Osteoarthritis usually occurs in joints that bear weight, such as the spine, knees, hips, and back. It is usually preceded by pain and symptoms of stiffness (often stiffness first, then pain), but swelling is not always present. In a small number of cases, osteoarthritis can cause disability. As the condition progresses, the bones can become more fragmented, increasing the likelihood of fractures. When osteoarthritis is more severe, bones can overgrow into osteophytes, known as bone spurs. These bone spurs can be detected with X-rays, usually near degenerative cartilage in the neck or waist. However, these changes typically do not alter the appearance of the affected area.

There are more than 28 types of peptides that make up collagen, with the more common types I, II, and III collagen accounting for about 90% of the total. Type II collagen forms joints. When collagen from pork bones and other sources is cooked at high temperatures, the collagen structure is destroyed, becoming denatured collagen. Additional supplements can only be used as general collagen and, therefore, cannot reduce the damage and inflammation of joint cartilage. Many studies have confirmed that the use of 'non-denatured type II collagen' (UC-II) can provide flexible maintenance for key parts. To achieve higher efficiency and longer-lasting effects, it is combined with glucosamine, chondroitin, and curcumin. In addition to providing resistance to compression in articular cartilage, it can also improve inflammation and significantly reduce pain in patients with primary osteoarthritis. Therefore, this research evaluated the effects of UCII, glucosamine and curcumin supplementation on knee pain and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Knee plain

Exclusion Criteria:

* Severe diseases of the heart, liver, kidneys, endocrine system, and other organs
* Long-term use of medication
* Infection, hypertension, diabetes, cerebrovascular disease, heart disease, liver disease, kidney disease, gastrointestinal disease
* Allergy to this product

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-12-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei medical university, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from social media between August 2024 and September 2024.
Pre-assignment Details: Of 32 enrolled participants, all of them met inclusion of criteria, but 2 of them were not included in the analysis because lost of follow-up.
Period: Overall Study
Arm/Group | Control Group | Test Group (UCII, Glucosamine, and Curcumin)
Started | 16 | 16
Completed | 15 | 15
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Test Group (UCII, Glucosamine, and Curcumin) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (16.65) | 34.8 (16.45) | 34.3 (16.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 15 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Points Change of Pain Evaluation Scale
Description: Self-assess pain using a visual analog scale (VAS), which is a straight line 10 cm in length, with 0 cm on the left representing no pain and 10 cm on the right representing extreme pain. Explain to the subjects that the pain intensity increases from left to right. Ask the subjects to mark the point on the line that corresponds to their pain level, and then record the distance in centimeters from the 0 cm mark.
  Record the points that the subjects wrote.
Time Frame: baseline, week 6, week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Test Group (UCII, Glucosamine, and Curcumin)
Number analyzed (Participants) | 15 | 15
score on a scale
  Normal walk, Left Baseline | 1.49 (1.19) | 1.15 (0.94)
  Normal walk, Left Week 6 | 1.15 (1.13) | 1.14 (1.08)
  Normal walk, Left Week 12 | 0.85 (1.05) | 0.50 (0.75)
  Normal walk, Right Baseline | 1.49 (1.19) | 1.15 (0.94)
  Normal walk, Right Week 6 | 1.29 (1.47) | 1.31 (1.10)
  Normal walk, Right Week 12 | 0.84 (1.00) | 0.63 (0.74)
  Stand up/squat down, Left Baseline | 2.83 (1.68) | 2.53 (1.61)
  Stand up/squat down, Left Week 6 | 1.81 (1.39) | 1.67 (1.22)
  Stand up/squat down, Left Week 12 | 1.29 (1.29) | 0.97 (0.85)
  Stand up/squat down, Right Baseline | 2.83 (1.68) | 2.53 (1.61)
  Stand up/squat down, Right Week 6 | 2.04 (1.72) | 1.78 (1.42)
  Stand up/squat down, Right Week 12 | 1.51 (1.35) | 1.20 (1.09)
  Bend to biggest angle, Left Baseline | 2.53 (2.22) | 1.50 (1.18)
  Bend to biggest angle, Left Week 6 | 1.54 (1.50) | 1.23 (1.47)
  Bend to biggest angle, Left Week 12 | 0.98 (1.12) | 0.52 (0.53)
  Bend to biggest angle, Right Baseline | 2.53 (2.22) | 1.50 (1.18)
  Bend to biggest angle, Right Week 6 | 1.54 (1.50) | 1.23 (1.47)
  Bend to biggest angle, Right Week 12 | 0.98 (1.12) | 0.52 (0.53)
Statistical Analysis 1: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); This analysis examined the overall (main) effect of treatment-comparing Control and Test groups across the three time points (baseline, week 6, and week 12) Comparison groups: Control and Test group of Normal walk, Left baseline, week 6, and week 12; Test type: Superiority; p = 0.478, ANOVA — It calculated the p value of two treatment (Control group and Test group). The threshold of statistical significance was p = 0.05
Statistical Analysis 2: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); This analysis examined the overall (main) effect of treatment-comparing Control and Test groups across the three time points (baseline, week 6, and week 12) Comparison groups: Control and Test group of Normal walk, Right baseline, week 6, and week 12; Test type: Superiority; p = 0.612, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); This analysis examined the overall (main) effect of treatment-comparing Control and Test groups across the three time points (baseline, week 6, and week 12) Comparison groups: Control and Test group of Stand up/squat down, Left baseline, week 6, and week 12; Test type: Superiority; p = 0.534, ANOVA
Statistical Analysis 4: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); This analysis examined the overall (main) effect of treatment-comparing Control and Test groups across the three time points (baseline, week 6, and week 12) Comparison groups: Control and Test group of Stand up/squat down, Right baseline, week 6, and week 12; Test type: Superiority; p = 0.538, ANOVA
Statistical Analysis 5: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); This analysis examined the overall (main) effect of treatment-comparing Control and Test groups across the three time points (baseline, week 6, and week 12) Comparison groups: Control and Test group of Bend to biggest angle, Left baseline, week 6, and week 12; Test type: Superiority; p = 0.195, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); This analysis examined the overall (main) effect of treatment-comparing Control and Test groups across the three time points (baseline, week 6, and week 12) Comparison groups: Control and Test group of Bend to biggest angle, Right baseline, week 6, and week 12; Test type: Superiority; p = 0.232, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); It calculated the interaction between 2 groups (Control group and Test group) X 3 time points (Baseline, week 6, week 12) of Normal walk, Left; Test type: Superiority; p = 0.369, ANOVA — It calculated the p value of the interaction between 2 groups X 3 time points. The threshold of statistical significance was p = 0.05
Statistical Analysis 8: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); It calculated the interaction between 2 groups (Control group and Test group) X 3 time points (Baseline, week 6, week 12) of Normal walk, Right; Test type: Superiority; p = 0.593, ANOVA — [p-value comment as in outcome 1, analysis 7]
Statistical Analysis 9: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); It calculated the interaction between 2 groups (Control group and Test group) X 3 time points (Baseline, week 6, week 12) of Stand up/squat down, Left; Test type: Superiority; p = 0.918, ANOVA — [p-value comment as in outcome 1, analysis 7]
Statistical Analysis 10: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); It calculated the interaction between 2 groups (Control group and Test group) X 3 time points (Baseline, week 6, week 12) of Stand up/squat down, Right; Test type: Superiority; p = 0.990, ANOVA — [p-value comment as in outcome 1, analysis 7]
Statistical Analysis 11: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); It calculated the interaction between 2 groups (Control group and Test group) X 3 time points (Baseline, week 6, week 12) of Bend to biggest angle, Left; Test type: Superiority; p = 0.263, ANOVA — [p-value comment as in outcome 1, analysis 7]
Statistical Analysis 12: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); It calculated the interaction between 2 groups (Control group and Test group) X 3 time points (Baseline, week 6, week 12) of Bend to biggest angle, Right; Test type: Superiority; p = 0.235, ANOVA — [p-value comment as in outcome 1, analysis 7]

2. Primary Outcome: Time Change of Up-and-go Test
Description: Timed up-and-go test (TUG) was a professional physical therapist marked a distance of 3 meters on the ground and placed an armless chair at one end. The subject sat on the chair with a straight back, and the time was measured from when the subject stood up and walked to the 3-meter mark at their usual speed, turned around, walked back, and sat down again. Shorter time spent indicates better knee function.
  Record the time that the subjects spent.
Time Frame: baseline, week 6, week 12
Measure: Mean (Standard Deviation); unit: unit of measure: seconds
Arm/Group | Control Group | Test Group (UCII, Glucosamine, and Curcumin)
Number analyzed (Participants) | 15 | 15
unit of measure: seconds
  Baseline | 9.96 (1.47) | 9.3 (0.98)
  Week 6 | 8.75 (0.68) | 8.83 (0.71)
  Week 12 | 8.64 (0.73) | 8.55 (0.76)
Statistical Analysis 1: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); This analysis examined the overall (main) effect of treatment-comparing Control and Test groups across the three time points (baseline, week 6, and week 12) Comparison groups: Control and Test group of up-and-go test on baseline, week 6, and week 12; Test type: Superiority; p = 0.399, ANOVA — [p-value comment as in outcome 1, analysis 1]; It calculated the p value of two treatment (Control group and Test group). The threshold of statistical significance was p = 0.05
Statistical Analysis 2: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); It calculated the interaction between 2 groups (Control group and Test group) X 3 time points (Baseline, week 6, week 12) of timed up-and-go test; Test type: Superiority; p = 0.106, ANOVA — [p-value comment as in outcome 1, analysis 7]

3. Primary Outcome: Degrees Change of Range of Motion (ROM)
Description: A professional physical therapist tested the active flexion and extension of the knee joint (range of motion, ROM) as the subjects attempted to achieve maximum active flexion and extension.
  Record the angle that the physical therapist measured. AROM: active range of motion; PROM: passive range of motion
Time Frame: baseline, week 6, week 12
Measure: Mean (Standard Deviation); unit: unit of measure: Degrees
Arm/Group | Control Group | Test Group (UCII, Glucosamine, and Curcumin)
Number analyzed (Participants) | 15 | 15
unit of measure: Degrees
  AROM, Left Baseline | 141.73 (6.84) | 137.67 (8.35)
  AROM, Left Week 6 | 141.20 (7.88) | 140.80 (8.54)
  AROM, Left Week 12 | 137.93 (7.66) | 136.80 (11.03)
  AROM, Right Baseline | 141.20 (6.70) | 138.00 (6.85)
  AROM, Right Week 6 | 140.80 (8.54) | 140.67 (8.57)
  AROM, Right Week 12 | 138.00 (7.78) | 138.67 (8.16)
  PROM, Left Baseline | 143.20 (7.08) | 139.33 (8.20)
  PROM, Left Week 6 | 143.07 (7.52) | 142.67 (8.27)
  PROM, Left Week 12 | 141.40 (7.67) | 138.80 (11.10)
  PROM, Right Baseline | 142.40 (6.60) | 139.73 (6.63)
  PROM, Right Week 6 | 142.67 (7.95) | 142.67 (8.30)
  PROM, Right Week 12 | 141.60 (7.14) | 140.13 (8.26)
Statistical Analysis 1: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); This analysis examined the overall (main) effect of treatment-comparing Control and Test groups across the three time points (baseline, week 6, and week 12) Comparison groups: Control and Test group of AROM, Left baseline, week 6, and week 12; Test type: Superiority; p = 0.502, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); This analysis examined the overall (main) effect of treatment-comparing Control and Test groups across the three time points (baseline, week 6, and week 12) Comparison groups: Control and Test group of AROM, Right baseline, week 6, and week 12; Test type: Superiority; p = 0.724, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); This analysis examined the overall (main) effect of treatment-comparing Control and Test groups across the three time points (baseline, week 6, and week 12) Comparison groups: Control and Test group of PROM, Left baseline, week 6, and week 12; Test type: Superiority; p = 0.414, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); This analysis examined the overall (main) effect of treatment-comparing Control and Test groups across the three time points (baseline, week 6, and week 12) Comparison groups: Control and Test group of PROM, Right baseline, week 6, and week 12; Test type: Superiority; p = 0.563, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); It calculated the interaction between 2 groups (Control group and Test group) X 3 time points (Baseline, week 6, week 12) of AROM, Left; Test type: Superiority; p = 0.110, ANOVA — [p-value comment as in outcome 1, analysis 7]
Statistical Analysis 6: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); It calculated the interaction between 2 groups (Control group and Test group) X 3 time points (Baseline, week 6, week 12) of AROM, Right; Test type: Superiority; p = 0.245, ANOVA — [p-value comment as in outcome 1, analysis 7]
Statistical Analysis 7: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); It calculated the interaction between 2 groups (Control group and Test group) X 3 time points (Baseline, week 6, week 12) of PROM, Left; Test type: Superiority; p = 0.113, ANOVA — [p-value comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); It calculated the interaction between 2 groups (Control group and Test group) X 3 time points (Baseline, week 6, week 12) of PROM, Right; Test type: Superiority; p = 0.395, ANOVA — [p-value comment as in outcome 1, analysis 7]

4. Primary Outcome: Points Change of Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), a widely used questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, and the total score was 96 points (Minimum: 0 points; Maximum: 96 points). The question content was divided into three parts: Pain (20 points), Stiffness (8 points), and Physical function (68 points). The higher score meant worse knee joint function.
  Record the points that the subjects got.
Time Frame: baseline, week 6, week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Test Group (UCII, Glucosamine, and Curcumin)
Number analyzed (Participants) | 15 | 15
score on a scale
  Pain Baeline | 5.73 (2.99) | 5.27 (2.52)
  Pain Week 6 | 4.47 (2.53) | 4.73 (2.94)
  Pain Week 12 | 4.07 (2.99) | 3.67 (2.72)
  Stiffness Baseline | 1.93 (1.39) | 1.60 (0.99)
  Stiffness Week 6 | 1.13 (0.92) | 1.53 (0.92)
  Stiffness Week 12 | 1.27 (1.22) | 1.33 (0.90)
  Physical function Baseline | 10.00 (8.64) | 9.00 (6.28)
  Physical function Week 6 | 6.47 (6.62) | 6.53 (4.76)
  Physical function Week 12 | 6.73 (8.56) | 4.87 (4.98)
Statistical Analysis 1: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); This analysis examined the overall (main) effect of treatment-comparing Control and Test groups across the three time points (baseline, week 6, and week 12) Comparison groups: Control and Test group of Pain on baseline, week 6, and week 12; Test type: Superiority; p = 0.823, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); This analysis examined the overall (main) effect of treatment-comparing Control and Test groups across the three time points (baseline, week 6, and week 12) Comparison groups: Control and Test group of Stiffness on baseline, week 6, and week 12; Test type: Superiority; p = 0.895, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); This analysis examined the overall (main) effect of treatment-comparing Control and Test groups across the three time points (baseline, week 6, and week 12) Comparison groups: Control and Test group of Physical function on baseline, week 6, and week 12; Test type: Superiority; p = 0.682, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); It calculated the interaction between 2 groups (Control group and Test group) X 3 time points (Baseline, week 6, week 12) of Pain; Test type: Superiority; p = 0.303, ANOVA — [p-value comment as in outcome 1, analysis 7]
Statistical Analysis 5: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); It calculated the interaction between 2 groups (Control group and Test group) X 3 time points (Baseline, week 6, week 12) of Stiffness; Test type: Superiority; p = 0.148, ANOVA — [p-value comment as in outcome 1, analysis 7]
Statistical Analysis 6: Comparison: Control Group vs Test Group (UCII, Glucosamine, and Curcumin); It calculated the interaction between 2 groups (Control group and Test group) X 3 time points (Baseline, week 6, week 12) of Physical function; Test type: Superiority; p = 0.283, ANOVA — [p-value comment as in outcome 1, analysis 7]

5. Primary Outcome: The Concentration of Serum Inflammatory Factors
Description: The concentration of interleukin-6 (IL-6), interleukin-1 beta (IL-1β), and tumor necrosis factor alpha (TNF-α) in serum.
Time Frame: baseline, week 6, week 12
Population: Data were not reported because the value was lower than limit of detection.
Measure: Mean (Standard Deviation); unit: unit of measure: concentration (pg/mL)
Arm/Group | Control Group | Test Group (UCII, Glucosamine, and Curcumin)
Number analyzed (Participants) | 15 | 15
unit of measure: concentration (pg/mL)
  IL-6 Baseline | NA (NA) — The data were below the lower limit of quantification. | NA (NA) — The data were below the lower limit of quantification.
  IL-6 Week 6 | NA (NA) — The data were below the lower limit of quantification. | NA (NA) — The data were below the lower limit of quantification.
  IL-6 Week 12 | NA (NA) — The data were below the lower limit of quantification. | NA (NA) — The data were below the lower limit of quantification.
  IL-1β Baseline | NA (NA) — The data were below the lower limit of quantification. | NA (NA) — The data were below the lower limit of quantification.
  IL-1β Week 6 | NA (NA) — The data were below the lower limit of quantification. | NA (NA) — The data were below the lower limit of quantification.
  IL-1β Week 12 | NA (NA) — The data were below the lower limit of quantification. | NA (NA) — The data were below the lower limit of quantification.
  TNF-α Baseline | NA (NA) — The data were below the lower limit of quantification. | NA (NA) — The data were below the lower limit of quantification.
  TNF-α Week 6 | NA (NA) — The data were below the lower limit of quantification. | NA (NA) — The data were below the lower limit of quantification.
  TNF-α Week 12 | NA (NA) — The data were below the lower limit of quantification. | NA (NA) — The data were below the lower limit of quantification.

ADVERSE EVENTS:
Time Frame: No applicable
Description: Death, serious adverse events, and others (non-serious adverse events) were not assessed for the study.
Arm/Group | Control Group | Test Group (UCII, Glucosamine, and Curcumin)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT06581094/Prot_SAP_000.pdf